CLINICAL TRIAL: NCT00015899
Title: Phase I Trial Of Escalating Oral Doses Of SCH 66336 In Pediatric Patients With Refractory Or Recurrent Brain Tumors
Brief Title: SCH 66336 in Treating Children With Recurrent or Progressive Brain Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pediatric Brain Tumor Consortium (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: James M. Boyett/PBTC Operations and Biostatistics Center Executive Director, Pediatric Brain Tumor Consortium
Purpose: Treatment
Other Study IDs: CDR0000068571; PBTC-003; SPRI-P02201
Record Dates: First submitted 2001-05-06; First posted 2003-01-27 (Estimated); Last update posted 2009-10-14 (Estimated); Status verified 2009-10

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: childhood craniopharyngioma; childhood central nervous system germ cell tumor; childhood oligodendroglioma; childhood choroid plexus tumor; childhood grade I meningioma; childhood grade II meningioma; childhood grade III meningioma; recurrent childhood cerebellar astrocytoma; recurrent childhood cerebral astrocytoma; recurrent childhood medulloblastoma; recurrent childhood visual pathway and hypothalamic glioma; recurrent childhood ependymoma; childhood atypical teratoid/rhabdoid tumor; childhood spinal cord neoplasm
MeSH Terms: conditions — Central Nervous System Neoplasms; Oligodendroglioma; Choroid Plexus Neoplasms; Astrocytoma; Medulloblastoma; Optic Nerve Glioma; Familial ependymoma; Rhabdoid Tumor; Spinal Cord Neoplasms | interventions — lonafarnib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: lonafarnib
  Other Names: SCH 66336

SUMMARY:
RATIONALE: SCH 66336 may stop the growth of tumor cells by blocking the enzymes necessary for cancer cell growth.

PURPOSE: This phase I trial is studying the side effects and best dose of SCH 66336 in treating children with recurrent or progressive brain tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the qualitative and quantitative toxicity of SCH 66336 in children with recurrent or progressive brain tumors.
* Estimate the maximum tolerated dose of this drug in these patients.
* Describe the pharmacokinetics of this drug with and without dexamethasone in these patients.
* Investigate the efficacy of this drug in these patients.

OUTLINE: This is a dose-escalation study.

Patients receive oral SCH 66336 twice daily. Treatment repeats every 4 weeks for a total of 26 courses in the absence of disease progression or unacceptable toxicity.

Cohorts of 1-6 patients receive escalating doses of SCH 66336 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose at which it is predicted that 20% of patients may experience dose-limiting toxicity. An additional 6 patients are treated at the determined MTD.

Patients are followed within 30 days of the last administration of the study drug and then for up to 3 months.

PROJECTED ACCRUAL: Approximately 25 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed recurrent or progressive (refractory) brain tumors

  * Histologic confirmation waived for brainstem gliomas
* Bone marrow involvement allowed if transfusion independent

PATIENT CHARACTERISTICS:

Age:

* 21 and under

Performance status:

* Lansky 60-100% OR
* Karnofsky 60-100%

Life expectancy:

* More than 8 weeks

Hematopoietic:

* See Disease Characteristics
* Absolute neutrophil count greater than 1,000/mm^3
* Platelet count greater than 75,000/mm^3
* Hemoglobin greater than 9 g/dL

Hepatic:

* Bilirubin no greater than upper limit of normal
* SGPT and SGOT less than 2.5 times normal
* Albumin greater than 3 g/dL
* PT/PTT no greater than 120% upper limit of normal
* No overt hepatic disease

Renal:

* Creatinine no greater than 1.5 times normal OR
* Glomerular filtration rate greater than 70 mL/min
* No overt renal disease

Cardiovascular:

* No overt cardiac disease

Pulmonary:

* No overt pulmonary disease

Other:

* Neurologic deficits allowed if stable for at least 1 week prior to study
* More than 3rd percentile weight for height
* Able to swallow pills
* No uncontrolled infection
* No known or suspected allergy to poloxamer 188, croscarmellose sodium, silicon dioxide, or magnesium stearate I
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for up to 10 weeks after study

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* More than 6 months since prior bone marrow transplantation
* More than 1 week since prior growth factors

Chemotherapy:

* At least 3 weeks since prior myelosuppressive chemotherapy (6 weeks for nitrosoureas) and recovered

Endocrine therapy:

* Concurrent dexamethasone allowed if on stable dose for at least 1 week prior to study
* Concurrent oral contraceptives or other hormonal contraceptive methods allowed

Radiotherapy:

* More than 6 weeks since prior substantial bone marrow radiotherapy
* More than 3 months since prior craniospinal radiotherapy (more than 24 Gy) or total body irradiation
* More than 2 weeks since prior focal radiotherapy for symptomatic metastatic sites

Surgery:

* Not specified

Other:

* No concurrent enzyme-inducing anticonvulsant drugs
* No other concurrent anticancer or experimental drug therapy

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 53 (Actual)
Dates: Start 2002-01; Primary Completion 2005-09 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Toxicities of SCH 66336 in children and adolescents with refractory CNS cancers
Maximum tolerated dose of SCH 66336 | Four weeks
Pharmacokinetics of SCH 66336

SECONDARY OUTCOMES:
Tumor response to SCH 66336

CONTACTS AND LOCATIONS:
Overall Officials: Mark W. Kieran, MD, PhD, Study Chair — Dana-Farber Cancer Institute
Locations (9):
- United States (9):
  - UCSF Comprehensive Cancer Center, San Francisco, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Texas Children's Cancer Center, Houston, Texas
  - Children's Hospital and Regional Medical Center - Seattle, Seattle, Washington

REFERENCES:
- [Result] Kieran MW, Packer RJ, Onar A, Blaney SM, Phillips P, Pollack IF, Geyer JR, Gururangan S, Banerjee A, Goldman S, Turner CD, Belasco JB, Broniscer A, Zhu Y, Frank E, Kirschmeier P, Statkevich P, Yver A, Boyett JM, Kun LE. Phase I and pharmacokinetic study of the oral farnesyltransferase inhibitor lonafarnib administered twice daily to pediatric patients with advanced central nervous system tumors using a modified continuous reassessment method: a Pediatric Brain Tumor Consortium Study. J Clin Oncol. 2007 Jul 20;25(21):3137-43. doi: 10.1200/JCO.2006.09.4243. PMID 17634493